CLINICAL TRIAL: NCT07064434
Title: Sacral Canal Block for Hip Replacement the Efficacy and Safety of Controlled Intraoperative Hypotension:a Single-center, Prospective, Randomized Controlled Study
Brief Title: Sacral Canal Block for Hip Replacement the Efficacy and Safety of Controlled Intraoperative Hypotension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wenxuan Ma-2025-1
Record Dates: First submitted 2025-05-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
Keywords: Sacral canal block; Hip replacement; Postoperative rehabilitation
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia group(NCB Group) (Active Comparator): Conventional general anesthesia was adopted, and laryngeal mask general anesthesia was only administered to the patient.
  Interventions: Procedure: Simple general anesthesia
- Sacral canal block + General anesthesia group (CB group) (Experimental): Thirty minutes before the start of the operation, 30ML of the pre-prepared 0.375% ropivacaine was injected into the sacral canal under ultrasound guidance, and the diffusion of the local anesthetic in the sacral canal could be observed.
  Interventions: Procedure: Sacral canal block combined with general anesthesia

INTERVENTIONS:
Procedure: Sacral canal block combined with general anesthesia — Sacral canal block: The patient lies on their side, with the back perpendicular to the edge of the operating table. The knee joints of the lower limbs are flexed, the thighs are close to the abdomen, and the waist is arched backward as much as possible, resembling a "shrimp" shape. The space between the sacrum and coccyx of the patient (sacral hiatus) is fully exposed. By using a low-frequency probe (such as 2-5 MHZ), the strong echo of the sacrum, the low echo of the sacral canal, and the echo of the surrounding soft tissues can be clearly seen. At the located sacral hiatus, hold the puncture needle and slowly insert it perpendicularly to the skin. When the puncture needle passes through the sacrococcygeal ligament, there will be a distinct "breakthrough sensation", which indicates that the puncture needle has entered the sacral canal. The general depth of needle insertion is about 2 to 3cm. However, the specific depth varies depending on factors such as the patient's body type.
  Arms: Sacral canal block + General anesthesia group (CB group)
Procedure: Simple general anesthesia — General anesthesia: Midazolam (0.2mg/kg), sufentanil (0.2-0.4μg/kg), etomidate (0.15-0.3 mg/kg), and rocuronium (0.6 mg/kg) were induced. After the patient's muscles were completely relaxed, a laryngeal mask was placed. Connect the anesthesia machine and set the ventilator parameters: Vol.Mode, tidal volume 6-8ml/kg, frequency 10-14 times /min, inhalation-exhalation ratio 1:2, and maintain EtCO2 at 35-45mmHg during the operation. Propofol (4-12mg/kg/h) and remifentanil (0.05-2ug/kg/min) were maintained. According to the operation course, rocuronium (0.15mg/kg) and sevoflurane inhalation (1% - 7%) could be administered at a single time. Anesthesiologists adjust the drug infusion rate based on the patient's hemodynamic indicators SBP, MAP, HR and clinical experience. When HR was less than 45 times /min during the operation, atropine was intravenously injected (0.25-0.5mg per time). When MAP is less than 55mmHg and lasts for more than 3 minutes, ephedrine (6-12mg each time) is given.
  Arms: General anesthesia group(NCB Group)

SUMMARY:
To observe the efficacy and safety of sacral canal block in controlled blood pressure reduction during hip replacement in the elderly, and to provide a better option for controlled blood pressure reduction during clinical hip surgery.

DETAILED DESCRIPTION:
Confirm the effectiveness of sacral canal block in controlled blood pressure reduction during hip replacement surgery in the elderly.

The patient underwent sacral canal block 30 minutes before the operation. The time from the start of the block to achieving the target blood pressure for controlled blood pressure reduction, the duration of the target blood pressure, and the blood pressure variability at different time points were observed. The blood pressure variability was used to evaluate the effect of controlled blood pressure reduction during the operation, the intraoperative blood loss, and the surgeon's satisfaction. It has been confirmed that sacral canal block can effectively achieve the purpose of controlled blood pressure reduction in hip replacement surgery for the elderly.

Clarify the safety of sacral canal block for controlled hypotension in hip replacement surgery.

The patient underwent sacral canal block 30 minutes before the operation. Observe from the start of the block to the regression of the block plane, and the patient was lowered Limb tissue oxygen saturation, peripheral perfusion index, unexpected hypotension, heart rate variability, pulse oxygen saturation, and whether there are complications related to sacral canal block such as local anesthetic poisoning, general spinal anesthesia, regional nerve injury, epidural hematoma, puncture site infection, etc. Meanwhile, the general information of the patients was recorded, including the duration of the operation, the consumption of opioids during the operation, the postoperative pain score, the incidence of nausea and vomiting, and the recovery of sensorimotor sensation in the postoperative block plane regression of the patients, etc. It is clear that sacral canal block can be safely used for controlled blood pressure reduction during hip replacement surgery in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Over 45 years old;
2. ASA Grade II - III;
3. BMI 18-35kg/㎡;
4. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Those who refuse to participate in the experiment;
2. Those who suffer from language or hearing impairments and are unable to communicate;
3. Those with contraindications for sacral canal block.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The onset time for blood pressure to drop from the basal blood pressure to the controlled antihypertensive target value | during surgery
  The onset time of blood pressure change from the basal blood pressure to the controlled blood pressure reduction target value (systolic blood pressure lower than or equal to 90mmHg or MAP60-70mmHg), the maintenance time of the target blood pressure value, the blood pressure values at each time point, and the intraoperative blood loss.

SECONDARY OUTCOMES:
Oxygen saturation of the lower extremity tissue on the healthy side（%） | during surgery
  Oxygen saturation of the lower extremity tissue on the healthy side（%）
Peripheral perfusion index | during surgery
  The peripheral perfusion index (PI) of the patients during the operation.
heart rate(times/minute) | during surgery
  The heart rate of the patients during the operation.
Intraoperative blood loss（Milliliters） | Day 1
  Compare the intraoperative blood loss of the two groups: Total blood loss = Total blood volume of the human body × (before Hct - after Hct)/average Hct.
The cumulative dosage of anesthetic drugs used | Day 1
  Compare the cumulative dosage of anesthetic drugs used during the operation in the two groups, whether other vasoactive drugs were used, and record the total fluid input volume during the operation in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No